CLINICAL TRIAL: NCT05796986
Title: Endovascular Treatment of Wide Neck Saccular Cerebral Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ayman Mohamed, Assistant lecturer of neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-03-02MD
Record Dates: First submitted 2023-03-14; First posted 2023-04-04 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Wide Neck Saccular Cerebral Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wide neck saccular cerebral aneurysms patients (Experimental)
  Interventions: Procedure: Endovascular procedure of treatment of wide neck saccular cerebral aneurysm

INTERVENTIONS:
Procedure: Endovascular procedure of treatment of wide neck saccular cerebral aneurysm — Endovascular different modalities for occlusion of wide neck saccular cerebral aneurysms include stent assisted coiling or balloon assisted coiling or flow diverter or 3D coiling

SUMMARY:
Intracranial aneurysm (IA) is a cerebrovascular disorder in which the weakness of a cerebral artery wall causes a localized dilation of the blood vessel. Intracranial aneurysm can develop and rupture, and about 85% of spontaneous subarachnoid hemorrhage (SAH) cases are caused by the rupture of Intracerebral aneurysm.

Two treatments are available globally: microsurgical clipping and endovascular treatment.

Endovascular treatment of Intracerebral aneurysms using detachable platinum coils ( was introduced in 1990 by Guido Guglielmi, an Italian neurosurgeon ) of different shapes and sizes are deposited into the aneurysm through a microcatheter, which reduces the blood flow and induces thrombus formation .

Wide neck aneurysm defined by neck diameter greater than 4 mm or dome-to-neck ratio less than 2 Despite advances in endovascular techniques , the treatment of wide-necked aneurysms remains problematic . Endovascular treatment of intracranial aneurysms is associated with lower morbidity and mortality rates and faster recovery compared with traditional microsurgical clipping.

In wide-necked Intracerebral aneurysms, complete coil embolization is often technically difficult owing to the risks of distal coil migration or coil impingement on the parent vessel .

Complete coil embolization using a single microcatheter without a supporting device in cases of wide-necked Intracerebral aneurysm is technically difficult. Total occlusion rates have increased recently as a result of the advancement of supporting devices These may include balloon remodeling, use of three-dimensional (3D) coils (Russian Doll Technique), combined use of stents and coils (Stent assisted coiling), flow diverters, use of intrasaccular flow disruption (like WEB), Double catheter Technique or combined extra- and intrasaccular devices.

ELIGIBILITY:
Inclusion Criteria:

* All patients of spontaneous subarachnoid haemorrhage due to ruptured wide neck saccular cerebral aneurysms
* unruptured Denovo wide neck saccular cerebral aneurysms

Exclusion Criteria:

* other forms of cerebral aneurysms rather than saccular type : fusiform and dissecting aneurysms
* complex aneurysms : giant and thrombosed aneyrsms
* any spontaneous subarachnoid haemorrhage with world fedriation of neurosurgery societies (WFNS) Grade 4&5
* Any patient unfit for general anesethia or has serious renal impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of procedure | 1 year
  degree of aneurysm occlusion classifeid by Raymond Roy classification

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Maher M, Schweizer TA, Macdonald RL. Treatment of Spontaneous Subarachnoid Hemorrhage: Guidelines and Gaps. Stroke. 2020 Apr;51(4):1326-1332. doi: 10.1161/STROKEAHA.119.025997. Epub 2020 Jan 22. No abstract available. PMID 31964292
- [Background] Lindgren A, Vergouwen MD, van der Schaaf I, Algra A, Wermer M, Clarke MJ, Rinkel GJ. Endovascular coiling versus neurosurgical clipping for people with aneurysmal subarachnoid haemorrhage. Cochrane Database Syst Rev. 2018 Aug 15;8(8):CD003085. doi: 10.1002/14651858.CD003085.pub3. PMID 30110521
- [Background] Kim JW, Park YS. Endovascular treatment of wide-necked intracranial aneurysms : techniques and outcomes in 15 patients. J Korean Neurosurg Soc. 2011 Feb;49(2):97-101. doi: 10.3340/jkns.2011.49.2.97. Epub 2011 Feb 28. PMID 21519497
- [Background] Pierot L, Wakhloo AK. Endovascular treatment of intracranial aneurysms: current status. Stroke. 2013 Jul;44(7):2046-54. doi: 10.1161/STROKEAHA.113.000733. No abstract available. PMID 23798560